CLINICAL TRIAL: NCT00499148
Title: Effect of Herbal Extract on Metabolic Parameters in Subjects With Type 2 Diabetes
Brief Title: Efficacy Study Testing Herbal Extract on Metabolic Parameters in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director, Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BJ82
Record Dates: First submitted 2007-07-05; First posted 2007-07-11 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: herbal extract; root of woody shrub grown in India/Sri-Lanka

SUMMARY:
The purpose of the study was to evaluate the effect of an herbal extract on postprandial glycemia following a meal.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* Between 18 and 75 years of age
* Male or non-pregnant, non-lactating female, at least 6 weeks postpartum
* If of childbearing potential, is practicing birth control
* BMI is more than or equal to 18kg/m2 and less than or equal to 35kg/m2
* If on anti-hyperglycemic, anti-hypertensive, lipid-lowering, or thyroid medications or hormone therapy, has been on constant dosage for at least 3 months prior to screening visit

Exclusion Criteria:

* Uses insulin for glucose control or has type 1 diabetes
* History of diabetic ketoacidosis.
* Current infection; surgery or corticosteroid treatment in the last 3 months or antibiotics in the last 3 weeks.
* Active malignancy
* Significant cardiovascular event less than or equal to 6 months prior to screening visit or history of congestive heart failure
* End state organ failure or status post organ transplant
* History of renal disease
* Current hepatic disease
* History of severe gastroparesis
* Has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV
* Currently taking herbals, dietary supplements, or medications, other than anti-hyperglycemic medications, during the past 4 weeks that could profoundly affect blood glucose
* Clotting or bleeding disorders
* Allergic or intolerant to any ingredient found in the study products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
positive AUC for plasma glucose | 4 hours

SECONDARY OUTCOMES:
positive AUC for serum insulin; adjusted peak values for plasma glucose and serum insulin; baseline plasma glucose and serum insulin concentrations; adjusted values for plasma glucose and serum insulin at individual postprandial time points. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A. Williams, MPH, Study Director — Abbott Nutrition
Locations (2):
- United States (2):
  - Radiant Research, Edina, Minnesota
  - Radiant Research, Cincinnati, Ohio